CLINICAL TRIAL: NCT02277002
Title: Reducing Commuter Air Pollutant Exposure by Cabin Air Filtration
Brief Title: Commuter Air Pollution Intervention Study
Acronym: CAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Canada (Other Government)
Responsible Party: Principal Investigator, Gary Mallach, Air Health Effects Researcher, Health Canada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: REB 2014-0006
Record Dates: First submitted 2014-10-09; First posted 2014-10-28 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Cognitive Function; Cardiopulmonary Function; Saliva Stress Hormones; Air Pollution Exposure; Lung Inflammation
Keywords: Cabin Air Filtration; Particulate Matter; Commuter Exposure; Traffic Related Air Pollution
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Placebo (Placebo Comparator): Participants are exposed to unfiltered cabin air
  Interventions: Other: Placebo
- Cabin Air Filter (Active Comparator): Participants are exposed to filtered cabin air
  Interventions: Device: Cabin Air Filtration

INTERVENTIONS:
Device: Cabin Air Filtration
  Arms: Cabin Air Filter
Other: Placebo — No Cabin Air Filtration
  Arms: Placebo

SUMMARY:
Traffic related air pollution is a well-recognised and much studied contributor to smog and is linked to a number of adverse health outcomes. Although traffic pollutants can travel long distances, exposure to the highest levels of the raw emissions can occur closest to the source; e.g. in a car in dense traffic conditions. Time spent in-vehicle may contribute up to half of commuters' daily exposure to certain air pollutants. Most new cars now have or allow for a cabin air filter, but it is not known how well cabin air filtration can reduce exposure to traffic-related air pollution.

This intervention study will measure commuters' exposure to air pollutants in rush hour traffic. It will evaluate the impact of this exposure on stress hormones in saliva, and short term cardiopulmonary health indicators such as blood pressure, heart rate variability and respiratory inflammation. It will also look at effects on cognition (mental processing and judgement) in this real world environment where any deficit could be important to safety. In addition, the study will examine whether cabin air filtration can reduce the exposure to traffic related air pollutants and result in improvements in short term cardiopulmonary and cognitive function. This research will contribute to our understanding of how this environment contributes to Canadians' overall air pollution exposure as well as the potential health impacts. It will also test a potentially valuable and economical means of reducing exposure to traffic related air pollution in a commuting environment. The study may also guide the future implementation of the use of cabin filters as an exposure reduction intervention.

Overall Project Objectives:

Can cabin air filtration effectively reduce exposure to traffic related air pollution? Does commuter exposure to air pollution affect short term stress, and cardiopulmonary and cognitive function? Can cabin air filtration mitigate the health effects of commuters' exposure to air pollution?

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals;
* non-smoking.

Exclusion Criteria:

* Smokers;
* living in a smoking household;
* currently experiencing seasonal allergies;
* suffering from heart rhythm problems or heart conditions;
* regularly taking corticosteroid medication;
* pregnant or breastfeeding;
* allergic to latex;
* sensitivity to adhesives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Variation in cardiopulmonary function | 5 hours
  Heart Rate Variability (HRV) will be measured from continuous ambulatory electrocardiogram (ECG) recordings collected during the study protocol. ECG will be worn for the duration of the study day period (approximately 5 hours), including a period prior to exposure and following exposure.

SECONDARY OUTCOMES:
Changes in neuropsychological Function | 5 hours
  Assessment of neuropsychological function can be achieved using a battery of mood and cognitive tests. The study will use a battery of tests that are comercially available through CANTAB, the mini-mental state exam designed by University of Cambridge. Battery will be administered before and after exposure.
Changes in endothelial function | 5 hours
  Endothelial function will be assessed using the non-invasive, FDA approved Endo-Pat2000 instrument. Test administration involves continuous measurement of blood flow and vascular tone in the fingertips of both index fingers, before, during and after an occlusion of blood flow to the non-dominant hand. Blood flow is occluded using a standard blood pressure cuff positioned on the upper arm. Measures will be carried out before and after exposure.
Changes in levels of Hypothalamic-Pituitary-Adrenal (HPA) Axis | 5 hours
  In the present study, salivary cortisol will be assessed as a non-invasive measure of HPA axis activation. Saliva sample collection will be done with Salivette swabs twice before exposure, once during exposure and twice following exposure.
Fraction of Exhaled Nitric Oxyde | 5 hours
  Lung inflammation will be assessed as the fraction of nitric oxide (NO) exhaled in the participants' breath using a portable, FDA approved, fractional exhaled nitric oxide (FENO) measurement device, the NIOX Mino. Measures will be carried out before and after exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Mallach, Principal Investigator — Health Canada
Locations (1):
- Guy-Favreau Complex, Montreal, Quebec, Canada